CLINICAL TRIAL: NCT01992757
Title: Comparison of Thromboelastography-derived Functional Fibrinogen Levels During and After Cardiopulmonary Bypass
Brief Title: Thromboelastography-derived Functional Fibrinogen Levels
Acronym: TEG-FF
Status: Completed | Type: Observational
Sponsor: University of Pennsylvania (Other)
Responsible Party: Sponsor
Other Study IDs: 818918
Record Dates: First submitted 2013-11-05; First posted 2013-11-25 (Estimated); Results first posted 2018-10-03 (Actual); Last update posted 2018-10-03 (Actual); Status verified 2017-11

CONDITIONS: Focus of Study; Coagulation Status of Cardiac Surgery Patient; Reducing Excess Blood Transfusion
Keywords: functional fibrinogen assay; cardiac surgery

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Cardiac surgery with cardiopulmary bypass

SUMMARY:
This study hopes to determine if thromboelastography-derived functional fibrinogen (TEG-FF or FLEV) levels obtained during the rewarming phase of cardiopulmonary bypass can provide information on coagulation status sooner, allowing for anticipation of post-bypass bleeding and transfusion requirements

ELIGIBILITY:
Inclusion Criteria:

* Elective cardiac surgery patients who are undergoing primary cardiac surgery

Exclusion Criteria:

* Emergency surgery
* Re-operative cardiac surgery
* History of hypercoagulable state as defined in medical record
* Anticoagulated status at time of surgery
* Plasma requirement prior to discontinuation of bypass (alters fibrinogen level)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The population for this study will be elective cardiac surgical patients who will be undergoing elective primary cardiac surgery.
Sampling Method: Non-Probability Sample
Enrollment: 51 (Actual)
Dates: Start 2013-11; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Prakash A Patel, MD, Principal Investigator — University of Pennsylvania Hospital
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Cardiac Surgery With Cardiopulmary Bypass: Patients over the age of 18 years undergoing cardiac surgery requiring CPB. Patients were excluded based on their need for emergency surgery, re-operative cardiac surgery, a history of coagulation disorders, and inability to sign consent.
Period: Overall Study
Arm/Group | Cardiac Surgery With Cardiopulmary Bypass
Started | 51
Completed | 49
Not Completed | 2
Not completed — 2 patients excluded due to FFP given. | 2

BASELINE CHARACTERISTICS:
Arm/Group | Cardiac Surgery With Cardiopulmary Bypass
Number analyzed (Participants) | 49
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 26
  >=65 years | 23
Age, Continuous [Mean (Full Range); unit: years] | 63.1 [22 to 84]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20
  Male | 29
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 49

OUTCOME MEASURES:

1. Primary Outcome: Change in Thromboelastography-derived Functional Fibrinogen Level (FLEV)
Description: FLEV values obtained during rewarming while on cardiopulmonary bypass (CPB) were compared to FLEV values obtained immediately after CPB and protamine administration. For all patients included, the mean values for rewarming FLEV and mean values for post-CPB FLEV were obtained. If the mean difference for the two timepoints was not statistically different by t-test, then the primary outcome would demonstrate the value of obtaining a rewarming FLEV sample.
Time Frame: Change in FLEV from rewarming and after cardiopulmonary bypass
Population: 49 patients undergoing cardiac surgery with CPB.
Measure: Mean (95% Confidence Interval); unit: mg/dL
Groups:
- FLEV Difference During Rewarming & Post-cardiopulmonary Bypass: All enrolled patients were in a single arm with multiple timepoints. FLEV values were obtained at baseline, rewarming, and post-CPB. The primary outcome was to compare the rewarming and post-CPB values to determine if a significant difference exists.
Arm/Group | FLEV Difference During Rewarming & Post-cardiopulmonary Bypass
Number analyzed (Participants) | 49
mg/dL | -1.1 [-25.8 to 23.6]

2. Secondary Outcome: Difference in Clauss Assay and FLEV
Description: This secondary outcome aimed to determine if standard laboratory assays for fibrinogen (Clauss) provided values similar to TEG-based functional fibrinogen (FLEV). The difference between the means at various timepoints is calculated in mg/dL.
Time Frame: Clauss vs FLEV for rewarming and post-CPB
Population: 49 patients undergoing cardiac surgery with CPB. The measure is the difference of the FLEV and the Clauss assay (i.e. FLEV minus Clauss since the FLEV is consistently higher).
Measure: Mean (95% Confidence Interval); unit: mg/dL
Groups:
- Clauss vs FLEV at Rewarming and Post-CPB: All enrolled patients were in a single arm with multiple timepoints. Clauss assay and FLEV values were obtained at baseline, rewarming, and post-CPB. The secondary outcome was to compare the rewarming and post-CPB values of Clauss value to FLEV to determine if a significant difference exists.
Arm/Group | Clauss vs FLEV at Rewarming and Post-CPB
Number analyzed (Participants) | 49
mg/dL
  Mean Clauss vs FLEV difference at rewarming | 120.6 [104.1 to 137.1]
  Mean Clauss vs FLEV difference post-CPB | 119.5 [101.7 to 137.4]

ADVERSE EVENTS:
Arm/Group | Cardiac Surgery With Cardiopulmary Bypass
All-Cause Mortality (participants affected / at risk) | 0/49
Serious Adverse Events (participants affected / at risk) | 0/49
Other Adverse Events (participants affected / at risk) | 0/49

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes